CLINICAL TRIAL: NCT01545726
Title: A Double-blind, Placebo-controlled Study Examining the Effect of Orally Administered QAW039 on Sputum Eosinophil Levels and Other Efficacy Outcomes in Patients With Sputum Eosinophilia and Persistent Asthma
Brief Title: Safety and Efficacy of QAW039 in Sputum Eosinophilia and Persistent Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQAW039A2208; 2011-004966-13 (EudraCT Number)
Record Dates: First submitted 2012-03-01; First posted 2012-03-07 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-10

CONDITIONS: Asthma
Keywords: Asthma; Sputum eosinophilia; CRTH2 receptor; PGD2 antagonist
MeSH Terms: conditions — Asthma | interventions — fevipiprant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- QAW039 (Experimental): Eligible patients will receive QAW039 po 450 mg daily dose.
  Interventions: Drug: QAW039
- Placebo (Placebo Comparator): Placebo to QAW039 (oral capsules) will be administered to match QAW039 schedule.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: QAW039 — QAW039 was supplied as capsules for oral administration.
  Arms: QAW039
Drug: Placebo — Placebo was supplied as capsules for oral administration.
  Arms: Placebo

SUMMARY:
This study will assess the safety and efficacy of QAW039 when added to current therapy in patients that have sputum eosinophilia and persistent asthma.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained before any assessment is performed.
2. Physician diagnosis of asthma, as per GINA guidelines GINA guidelines and currently prescribed ICS or ICS-LABA therapy.
3. Patients who are demonstrated to have reversible airway obstruction, significant FEV1 variability or airway hyperresponsiveness (AHR), or who have shown such responses in previous test(s) within the last five years.
4. An ACQ score ≥ 1.5 at randomization or ≥ 1 exacerbations (requiring higher than the patient's normal dose of OCS or IV corticosteroids for ≥ 3 days) in the past 12 months. The definition of exacerbations includes episodes during which the patient self-administered higher doses of OCS as part of a documented self-management plan initiated by the patient's general practitioner or respiratory physician.
5. Patients currently on GINA step 2 to step 5 asthma therapies.
6. Sputum eosinophil count ≥ 2% at screening.

Exclusion Criteria:

1. Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer.
2. History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes (CRTH2 antagonists).
3. History of long QT syndrome or whose QTc interval (Fridericia's) is prolonged >450 msec for males and >470 msec for females at screening or baseline.
4. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
5. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (> 5 mIU/mL).
6. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using effective methods of contraception during the study treatment and for 5 days (5 half-lives) after treatment.
7. Acute illness other than asthma which, in the investigator's opinion, may compromise the well-being of the patient or study endpoint assessments at the start of the study
8. Patients who are considered unsuitable for inclusion by the assessing physician due to serious co-morbidities such as cancer, emphysema or significant bronchiectasis.
9. Recent (within 6 weeks of screening) or current lower respiratory tract infection.
10. Patients who have been hospitalized or required high-dose (>10mg prednisolone/day) oral corticosteroid (OCS) therapy within 6 weeks of the screening visit.
11. Patients with clinically significant laboratory abnormalities (not associated with the study indication) at screening.
12. Patients who have a clinically significant abnormality on a 12-lead ECG recorded within one month prior to or at screening.
13. Patients with a body mass index (BMI) < 17 or > 40 kg/m2.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2012-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in sputum eosinophil percentage at week 12 (baseline measurement is defined as sputum eosinophil percentage at Day1 prior to the first dosing). | Visit 3 (day 1); Visit 5 (day 84)
  Sputum induction is performed through the inhalation of hypertonic saline. Sputum is collected and assessed for differential cellular content (absolute numbers and percentages). The primary variable will be summarized by treatment and analyzed using an ANCOVA model with treatment as the fixed effect and the respective baseline value as the covariate.

SECONDARY OUTCOMES:
Change from baseline to week 12 in Asthma Control Questionnaire (ACQ) | Visit 3 (day 1); Visit 5 (day 84)
  Participants complete the Asthma Control Questionnaire (ACQ). The ACQ has 7 equally weighted items; 5 on symptom assessment, 1 on rescue bronchodilator use and 1 on airway caliber Forced Expiratory Volume in one second (FEV1) % predicted. Items 1-6 are scored along a 7 point response scale, where 0 = good control and 6 = poor control. The 7th item on % predicted FEV1 (pre-bronchodilator) is scored by clinic staff on a 7 point scale. Secondary variables are summarized by treatment and analyzed using ANCOVA model with treatment as the fixed effect and the respective baseline value as covariate.
Safety and tolerability of QAW039 in patients with moderate to severe asthma | Visit 2 (day -14); Visit 3 (day 1); Visit 4 (day 42); Visit 5 (day 84); Visit 6 (day 126)
  All safety endpoints (including adverse events, laboratory data, vital signs and ECG) will be summarized by treatment group for all patients in the safety population. All data will be included in the analysis regardless of rescue medication use.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Leicester, United Kingdom

REFERENCES:
- [Derived] Gonem S, Berair R, Singapuri A, Hartley R, Laurencin MFM, Bacher G, Holzhauer B, Bourne M, Mistry V, Pavord ID, Mansur AH, Wardlaw AJ, Siddiqui SH, Kay RA, Brightling CE. Fevipiprant, a prostaglandin D2 receptor 2 antagonist, in patients with persistent eosinophilic asthma: a single-centre, randomised, double-blind, parallel-group, placebo-controlled trial. Lancet Respir Med. 2016 Sep;4(9):699-707. doi: 10.1016/S2213-2600(16)30179-5. Epub 2016 Aug 5. PMID 27503237